CLINICAL TRIAL: NCT03984851
Title: Hemostasis Using Surgicel in Pediatric Tonsillectomy
Status: Completed | Type: Observational
Sponsor: Dr. Abdul Mohsen Ibrahim Al-Turki Clinic (Other)
Responsible Party: Principal Investigator, Abdulmohsen Al-Terki, Dr. Abdulmohsen Al-Terki, Dr. Abdul Mohsen Ibrahim Al-Turki Clinic
Other Study IDs: Al-Terki Clinic
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Tonsil; Injury; Surgical Blood Loss
Keywords: tonsillectomy; primary hemostasis tonsillectomy; surgicel
MeSH Terms: conditions — Wounds and Injuries; Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: Surgicel Group: a retrospective cohort study. Two groups were assigned, the first under the care of the author [AA], in which patients of his group underwent cold dissection tonsillectomy and achieved hemostasis via surgicel (without bipolar cautery). While group B patients (consisted of 2 surgeons) underwent cold dissection tonsillectomy and attained hemostasis with bipolar cautery. The main outcome that was pursued was postoperative tonsillectomy bleeding
- Group B: Bipolar Cautery group: a retrospective cohort study. Two groups were assigned, the first under the care of the author [AA], in which patients of his group underwent cold dissection tonsillectomy and achieved hemostasis via surgicel (without bipolar cautery). While group B patients (consisted of 2 surgeons) underwent cold dissection tonsillectomy and attained hemostasis with bipolar cautery. The main outcome that was pursued was postoperative tonsillectomy bleeding

SUMMARY:
Tonsillectomy is one of the commonest procedures performed in otolaryngology and one of its major complications is post-tonsillectomy bleeding.

The goal of this study was to assess the effectiveness of Surgicel without bipolar cautery in achieving primary hemostasis in tonsillectomy. The patient that were enrolled in this retrospective study were patients who underwent tonsillectomy and achieved hemostasis either by Surgicel (group A) or bipolar cautery (group B). Our results showed that there was no statistical significant difference between the two techniques in terms of post-operative bleeding events.

DETAILED DESCRIPTION:
Tonsillectomy is one of the commonest procedures performed in otolaryngology and one of its major complications is post-tonsillectomy bleeding.

The goal of this study was to assess the effectiveness of Surgicel without bipolar cautery in achieving primary hemostasis in tonsillectomy.

The study was a retrospective cohort in three tertiary care centers in xxxx, from January 2016 to August 2018. All patients underwent at least tonsillectomy, with a proportion undergoing additional adenoidectomy, myringotomy, or tube insertion as indicated, were enrolled in the study. Patients were stratified to 2 groups according to the surgeons preference for the hemostasis technique, one was subjected to cold dissection tonsillectomy and achieved hemostasis via the application of Surgicel to the surgical site, and the other underwent cold dissection tonsillectomy and attained hemostasis through bipolar cautery.

ELIGIBILITY:
Inclusion Criteria:

* Patients under age of 12, diagnosed with recurrent tonsillitis or OSA and are candidates for tonsillectomy
* patients must have went tonsillectomy

Exclusion Criteria:

* age more than 12

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: any patient under the age of 12 who underwent tonsillectomy due to either recurrent tonsillitis or OSA by the 3 consultant otolaryngology surgeon authors in the study
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Primary Post-operative tonsillectomy bleeding | 24 hours post-op
  Bleeding due to the surgical procedure within 24 hours from the surgery
Secondary Post-operative Tonsillectomy bleeding | after 24 hours
  Bleeding due to the surgical procedure after 24 hours from the surgery

IPD SHARING:
Plan to Share IPD: Undecided